CLINICAL TRIAL: NCT02343042
Title: A Phase 1b/2 Study of Selinexor (KPT-330) in Combination With Backbone Treatments for Relapsed/Refractory Multiple Myeloma and Newly Diagnosed Multiple Myeloma
Brief Title: Selinexor and Backbone Treatments of Multiple Myeloma Patients
Acronym: STOMP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-017
Record Dates: First submitted 2015-01-13; First posted 2015-01-21 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Selinexor; KCP-330; STOMP; Multiple Myeloma; Relapsed/Refractory; Dexamethasone; Pomalidomide; Bortezomib; Karyopharm; Lenalidomide; Daratumumab; Newly Diagnosed; Carfilzomib; Ixazomib; Elotuzumab; Clarithromycin; Belantamab mafodotin; Mezigdomide; CC-92480; BMS-986348
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — selinexor; Dexamethasone; Calcium Dobesilate; Lenalidomide; pomalidomide; Bortezomib; daratumumab; carfilzomib; ixazomib; elotuzumab; Clarithromycin; belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- 1: Selinexor, Low-dose Dexamethasone and Pomalidomide (SPd) (Experimental): Each cycle is of 28 days
  Cohort 1.1: Selinexor (SEL) 60/80/100 mg orally (PO) once weekly (QW); Dexamethasone (DEX) 40 mg PO once weekly; Pomalidomide (POM) 2/3/4 mg PO Days 1-21.
  Cohort 1.2: SEL 40/60/80 mg PO twice weekly (BIW); DEX 20 mg PO twice weekly; POM 3/4 mg PO Days 1-21.
  Cohort 1.3: Selinexor, Dexamethasone and Pomalidomide will be dosed at RP2D-1.
  Cohort 1.4: SEL 40 mg PO QW; DEX 40 mg PO QW; POM 4mg PO once daily (QD) Days 1-21.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Pomalidomide
- 2: Selinexor, Low-dose Dexamethasone and Bortezomib (SVd) (Experimental): Each cycle is of 35 days
  Cohort 2.1: SEL 60/80/100 mg PO once weekly; DEX 40 mg PO once weekly; Bortezomib (BOR) 1.3 milligram per meter square (mg/m^2) subcutaneous (SC) once weekly.
  Cohort 2.2: SEL 40/60/80 mg PO twice weekly; DEX 20 mg PO twice weekly; BOR 1.3 mg/m^2 subcutaneous (SC) once weekly.
  Cohort 2.3: Selinexor, Dexamethasone and Bortezomib will be dosed at RP2D-2.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Bortezomib
- 3: Selinexor, Low-dose DEX, and Lenalidomide (SRd) in RRMM (Experimental): Each cycle is of 28 days
  Cohort 3.1: SEL 40/60/80/100 mg PO once weekly; DEX 40 mg PO once weekly; Lenalidomide (LEN) 15/25 mg PO Days 1-21.
  Cohort 3.2: SEL 40/60/80 mg PO twice weekly; DEX 20 mg PO twice weekly; LEN 15/25 mg PO Days 1-21.
  Cohort 3.3: Selinexor, Dexamethasone and Lenalidomide will be dosed at RP2D-3.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Lenalidomide
- 4:Selinexor, Low-dose dexamethasone, Pomalidomide, Velcade (SPVd) (Experimental): PK Run-in Period: Selinexor and Clarithromycin:
  * For the first 9 patients enrolled into this dose escalation arm
  * 14 day run-in period after which patients will proceed to Dose-Escalation Phase C1D1
  Selinexor 40 mg will be dosed on Days 1 and 8. Clarithromycin 500 mg will be dosed twice daily on Days 2-8.
  PK samples will be collected on Days 1 and 8 at 1, 1.5, 2, 3, 4, 5, 6, 8, and 24 hours post dose.
  Dose-escalation Phase:
  * All patients enrolled into this Arm
  * Each cycle is of 28 days.
  Cohort 4.1:
  SEL 40/60 mg PO once weekly; DEX 40 mg PO once weekly; POM 4 mg PO Days 1-21; BOR 1.3 mg/m^2 subcutaneous (SC) once weekly.
  Cohort 4.3: Selinexor, Dexamethasone, Pomalidomide, Velcade (Bortezomib) will be dosed at RP2D-4.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Pomalidomide; Drug: Bortezomib; Drug: Clarithromycin
- 5: Selinexor, Low-dose dexamethasone, and Daratumumab (SDd) (Experimental): Each cycle is of 28 days
  Cohort 5.1:
  SEL 80/100 mg PO once weekly; DEX 40 mg once weekly (IV or PO); DARA: 16 mg/kg IV infusion Cycle 1-2: Once weekly, Cycle 3-6: Every other week, Cycle 6 and greater: Once a month.
  Cohort 5.2:
  SEL: 60 mg PO twice weekly; DEX: 40 mg weekly (IV or PO); DARA: 16 milligram per kilogram (mg/kg) IV infusion Cycle 1-2: Once. weekly, Cycle 3-6: Every other week, Cycle 6 and greater: Once a month.
  Cohort 5.3: Selinexor, Dexamethasone and Daratumumab will be dosed at RP2D-5.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Daratumumab
- 6: Selinexor, Low-dose dexamethasone, and Carfilzomib (SKd) (Experimental): PK Run-in Period: Selinexor and Clarithromycin:
  * For the first 9 patients enrolled into this dose escalation arm
  * 14 day run-in period after which patient will proceed to Dose-Escalation Phase C1D1
  Selinexor 40 mg will be dosed on Days 1 and 8. Clarithromycin 500 mg will be dosed twice daily on Days 2-8.
  PK samples will be collected on Days 1 and 8 at 1, 1.5, 2, 3, 4, 5, 6, 8, and 24 hours post dose.
  Dose-Escalation Phase:
  * All patients enrolled into this Arm
  * Each cycle is of 28 days
  Cohort 6.1:
  SEL 40/60/80/100 mg PO once weekly on days 1, 8, 15, and 22; DEX 40 mg IV or PO once weekly; Carfilzomib (CAR) 56 or 70 mg/m^2 IV infusion once weekly on days 1, 8, and 15.
  Cohort 6.2:
  SEL 60/80/100 mg PO once weekly on days 1, 8, and 15; DEX 40 mg IV or PO once weekly; CAR 56 or 70 mg/m^2 IV infusion once weekly on days 1, 8, and 15.
  Cohort 6.3: Selinexor, Dexamethasone and Carfilzomib will be dosed at RP2D-6.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Carfilzomib; Drug: Clarithromycin
- 7: Selinexor, Low-dose DEX and Lenalidomide (SRd) in NDMM (Experimental): Each cycle is of 28 days
  Cohort 7.1:
  SEL 40/60/80 mg PO once weekly; DEX 40 mg PO once weekly; LEN 25 mg PO Days 1-21.
  Cohort 7.3: Selinexor, Dexamethasone and Lenalidomide will be dosed at RP2D-7.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Lenalidomide
- 8: Selinexor, Low-dose dexamethasone, and Ixazomib (SNd) (Experimental): PK Run-in Period: Selinexor & Clarithromycin:
  * For the first 9 patients enrolled into this dose escalation arm
  * 14 day run-in period after which patient will proceed to Dose-Escalation Phase C1D1
  Selinexor 40 mg will be dosed on Days 1 and 8. Clarithromycin 500 mg will be dosed twice daily on Days 2-8.
  PK samples will be collected on Days 1 and 8 at 1, 1.5, 2, 3, 4, 5, 6, 8, and 24 hours post dose.
  Dose-Escalation Phase:
  * All patients enrolled into this Arm
  * Each cycle is of 28 days
  Cohort 8.1:
  SEL 40/60/80/100 mg PO once weekly; DEX 20 mg PO twice weekly; IXA 3/4 mg PO once weekly.
  Cohort 8.3: Selinexor, Dexamethasone and Ixazomib will be dosed at RP2D-8.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Ixazomib; Drug: Clarithromycin
- 9: Selinexor, Low-dose DEX, Pomalidomide and Elotuzumab (SPEd) (Experimental): PK Run-in Period: Selinexor and Clarithromycin:
  * For the first 9 patients enrolled into this dose escalation arm
  * 14 day run-in period after which patient will proceed to Dose-Escalation Phase C1D1
  Selinexor 40 mg will be dosed on Days 1 and 8. Clarithromycin 500 mg will be dosed twice daily on Days 2-8.
  PK samples will be collected on Days 1 and 8 at 1, 1.5, 2, 3, 4, 5, 6, 8, and 24 hours post dose.
  Dose-Escalation Phase:
  * All patients enrolled into this Arm
  * Each cycle is of 28 days
  Cohort 9.1:
  SEL 20/40/60 mg PO once weekly; DEX 28/20 mg PO twice weekly; POM 4 mg PO QD Days 1-21; Elotuzumab (ELO) 10/20 mg/kg IV will be given once weekly on Days 1,8, 15 and 22 of Cycles 1-2. Starting on Cycle 3 and continuing for future cycles, elotuzumab will be dosed at 20 mg/kg on Day 1 of each cycle only.
  Cohort 9.3: Selinexor, Dexamethasone, Pomalidomide and Elotuzumab will be dosed at RP2D-9.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Pomalidomide; Drug: Elotuzumab
- 10. Selinexor, Dexamethasone, and Belantamab Mafodotin (SBd) (Experimental): Each cycle is of 21 days
  Cohort 10.1:
  SEL 40/60/80 mg PO once weekly on Days 1, 8, and 15; DEX 40 mg PO QW on Days 1, 8, and 15; Belantamab Mafodotin (BEL) 2.5 mg/kg IV infusion every 3 weeks (Q3W) Day 1 of each cycle.
  Cohort 10.3:
  Selinexor, Dexamethasone, and Belantamab Mafodotin will be dosed at RP2D-10.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Belantamab Mafodotin
- 11. Selinexor, Dexamethasone, Pomalidomide, and Daratumumab (SDPd) (Experimental): Each Cycle is of 28 days
  Cohort 11.1 SEL 40/60 mg PO once weekly on Days 1, 8, and 15; DEX total 40 mg weekly (IV or PO) single or divided doses on Days 1, 8, 15, and 22; POM 4 mg PO QW Days 1-21; DARA 16 mg/kg IV or SC QW on Days 1, 8, 15 and 22 of Cycles 1-2 and on Days 1 and 15 of Cycles 3-6, Day 1 of every Cycle greater than (>6).
  Cohort 11.3 Selinexor, Dexamethasone, Pomalidomide, and Daratumumab will be dosed at RP2D-11.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Pomalidomide; Drug: Daratumumab
- 12. Selinexor + dexamethasone + mezigdomide (SMd) (Experimental): The dose of selinexor will be formally escalated from 40 mg QW to 60 mg QW in combination with mezigdomide 0.6 mg daily. Mezigdomide dosing may be de-escalated as per 3+3 criteria to 0.3 mg or escalated to 1.0 mg. The dose level that passes DLT evaluation will be considered the MTD for the cohort.
  Interventions: Drug: Selinexor; Drug: Dexamethasone; Drug: Mezigdomide

INTERVENTIONS:
Drug: Selinexor — Oral tablets
  Other Names: KPT-330; XPOVIO®
Drug: Dexamethasone — Oral tablets
  Other Names: Decadron®
Drug: Lenalidomide — Oral capsule
  Other Names: Revlimid®
  Arms: 3: Selinexor, Low-dose DEX, and Lenalidomide (SRd) in RRMM; 7: Selinexor, Low-dose DEX and Lenalidomide (SRd) in NDMM
Drug: Pomalidomide — Oral tablets
  Other Names: Pomalyst®
  Arms: 11. Selinexor, Dexamethasone, Pomalidomide, and Daratumumab (SDPd); 1: Selinexor, Low-dose Dexamethasone and Pomalidomide (SPd); 4:Selinexor, Low-dose dexamethasone, Pomalidomide, Velcade (SPVd); 9: Selinexor, Low-dose DEX, Pomalidomide and Elotuzumab (SPEd)
Drug: Bortezomib — Subcutaneous Injection (single use vial)
  Other Names: Velcade®
  Arms: 2: Selinexor, Low-dose Dexamethasone and Bortezomib (SVd); 4:Selinexor, Low-dose dexamethasone, Pomalidomide, Velcade (SPVd)
Drug: Daratumumab — Intravenous Infusion
  Other Names: Darzalex®
  Arms: 11. Selinexor, Dexamethasone, Pomalidomide, and Daratumumab (SDPd); 5: Selinexor, Low-dose dexamethasone, and Daratumumab (SDd)
Drug: Carfilzomib — Intravenous infusion
  Other Names: Kyprolis®
  Arms: 6: Selinexor, Low-dose dexamethasone, and Carfilzomib (SKd)
Drug: Ixazomib — Oral capsule
  Other Names: Ninlaro®
  Arms: 8: Selinexor, Low-dose dexamethasone, and Ixazomib (SNd)
Drug: Elotuzumab — Intravenous infusion
  Other Names: Empliciti®
  Arms: 9: Selinexor, Low-dose DEX, Pomalidomide and Elotuzumab (SPEd)
Drug: Clarithromycin — Tablets
  Other Names: Biaxin
  Arms: 4:Selinexor, Low-dose dexamethasone, Pomalidomide, Velcade (SPVd); 6: Selinexor, Low-dose dexamethasone, and Carfilzomib (SKd); 8: Selinexor, Low-dose dexamethasone, and Ixazomib (SNd)
Drug: Belantamab Mafodotin — Intravenous infusion
  Other Names: BLENREP
  Arms: 10. Selinexor, Dexamethasone, and Belantamab Mafodotin (SBd)
Drug: Mezigdomide — Oral Capsules
  Other Names: BMS-986348; CC-92480
  Arms: 12. Selinexor + dexamethasone + mezigdomide (SMd)

SUMMARY:
This study will independently assess the efficacy and safety of 11 combination therapies in 12 arms, in dose-escalation/-evaluation and expansion phases, for the treatment of patients with relapsed/refractory multiple myeloma (RRMM) and newly diagnosed multiple myeloma (NDMM). The combinations to be evaluated are:

* Arm 1: Selinexor + dexamethasone + pomalidomide (SPd); enrollment complete
* Arm 2: Selinexor + dexamethasone + bortezomib (SVd); enrollment complete
* Arm 3: Selinexor + dexamethasone + lenalidomide (SRd) in RRMM; enrollment complete
* Arm 4: Selinexor + dexamethasone + pomalidomide + bortezomib (SPVd); enrollment complete
* Arm 5: Selinexor + dexamethasone + daratumumab (SDd); enrollment complete
* Arm 6: Selinexor + dexamethasone + carfilzomib (SKd); enrollment complete
* Arm 7: Selinexor + dexamethasone + lenalidomide (SRd) in NDMM; enrollment complete
* Arm 8: Selinexor + dexamethasone + ixazomib (SNd); enrollment complete
* Arm 9: Selinexor + dexamethasone + pomalidomide + elotuzumab (SPEd); enrollment complete
* Arm 10: Selinexor + dexamethasone + belantamab mafodotin (SBd); enrollment complete
* Arm 11: Selinexor + dexamethasone + pomalidomide + daratumumab (SDPd); enrollment complete
* Arm 12: Selinexor + dexamethasone + mezigdomide (SMd); actively recruiting

Selinexor pharmacokinetics:

* PK Run-in (Days 1-14):

Starting in protocol version 8.0, patients enrolled to any arm in the Dose Escalation Phase (i.e., Arm 4 [SPVd], Arm 6 [SKd], Arm 8 [SNd], Arm 9 [SPEd], Arm 10 [SBd], and Arm 11 [SDPd]) will also first be enrolled to a pharmacokinetics (PK) Run-in period until 9 patients have been enrolled to this period to evaluate the PK of selinexor before and after co-administration with a strong CYP3A4 inhibitor. This run-in period does not apply to Arm 12 (SMd).

DETAILED DESCRIPTION:
This is a multi-center, open-label, clinical study with Dose Escalation (Phase 1) and Expansion (Phase 2) to independently assess the MTD, efficacy , and safety of 11 combination therapies in 12 arms in patients with RRMM and NDMM. Patients will be assigned to treatment arms based on their diagnoses and treatment histories. For 9 patients, a PK Run-in period will precede Cycle 1 (DLT evaluation) to assess selinexor PK when co-administered with a strong CYP3A4 inhibitor. In the Dose Escalation Phase (Phase 1): (a) in Arm 1 (SPd), Arm 2 (SVd), and Arm 3 (SRd in RRMM), patients will be randomized to either QW or BIW selinexor dosing cohorts; (b) in Arm 5 (SDd), patients will be sequentially assigned in blocks of 3 to either QW or BIW selinexor dosing; (c) in Arm 4 (SPVd), Arm 6 (SKd), Arm 7 (Srd in NDMM), Arm 8 (SNd), Arm 9 (SPEd), Arm 10 (SBd), Arm 11 (SDPd), and Arm 12 (SMd) patients will be assigned to QW selinexor dosing.

Cohort 1.4 is included from Version 10 to study safety and tolerability of SPd with selinexor 40 mg QW, is lower than RP2D (ie, selinexor 60 mg QW) in combination with pomalidomide 4 mg. Cohort 1.4 is a different expansion cohort from the one with RP2D (ie, Cohort 1.3). In Cohort 1.4, 20 patients will be enrolled in total.

Starting in protocol Version 8.0, patients enrolled to the Dose Escalation Phase of Arm 4 (SPVd), Arm 6 (SKd), Arm 8 (SNd), Arm 9 (SPEd), Arm 10 (SBd), and Arm 11 (SDPd) will first be enrolled to a 14-day PK Run-in period (selinexor +/- clarithromycin) until 9 patients have been enrolled. During this 14-day PK Run-in period, selinexor 40 milligrams (mg) will be administered alone on Day 1, clarithromycin 500 mg twice daily (BID) will be administered on Days 2-8, and selinexor 40 mg will again be administered on Day 8 with the morning clarithromycin dose. Blood samples for PK analysis will be collected pre-dose and 1 (± 10 min), 1.5 (± 10 min), 2 (± 10 min), 3 (± 10 min), 4 (± 10 min), 5 (± 10 min), 6 (± 10 min), 8 (± 10 min), and 24 h (± 30 min) hours after selinexor is dosed on Day 1 (without clarithromycin) and Day 8 (with clarithromycin). Patients will then proceed to the DLT evaluation period that will begin after the completion of the 14-day PK Run-in period; this day will be designated as Cycle 1 Day 1 (C1D1) in the Dose Escalation Phase.

Starting in protocol v12, in Arm 12 (SMd) additional PK sampling for mezigdomide will be collected concurrently with selinexor on Cycle 1 Day 1 (C1D1) at 2,4, and 6 hrs post-mezigdomide/selinexor dose; additional mezigdomide PK samples will be collected pre-mezigdomide dose on Days 8 and 15 of Cycles 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed in accordance with federal, local, and institutional guidelines.
2. Age greater than or equal to (≥) 18 years at the time of informed consent.
3. Histologically confirmed diagnosis with measurable disease for relapsed/refractory myeloma.
4. Symptomatic MM, based on IMWG guidelines.
5. Patients must have measurable disease as defined by at least one of the following:

   1. Serum M-protein ≥ 0.5 gram per deciliter (g/dL) by serum protein electrophoresis (SPEP) or, for immunoglobulin A (IgA) myeloma, by quantitative IgA
   2. Urinary M-protein excretion at least 200 mg/24 hours
   3. Serum free light chain (FLC) ≥ 100 milligram per liter (mg/L), provided that FLC ratio is abnormal
   4. If SPEP is felt to be unreliable for routine M-protein measurement (example, for IgA MM), then quantitative immunoglobulin (Ig) levels by nephelometry or turbidometry are acceptable
6. Any non-hematological toxicities (except for peripheral neuropathy as described in exclusion criterion #22) that patients had from treatments in previous clinical studies must have resolved to less than or equal (≤) Grade 2 by C1D1.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
8. Adequate hepatic function within 28 days prior to C1D1:

   * For SPd, SRd, and SPEd: Total bilirubin < 2* upper limit of normal (ULN) (except patients with Gilbert's syndrome [hereditary indirect hyperbilirubinemia] who must have a total bilirubin of ≤ 3* ULN) and both aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5* ULN
   * For SVd, SPVd, SDd, SNd, SBd and SDPd: Total bilirubin of < 1.5* ULN (except patients with Gilbert's syndrome [hereditary indirect hyperbilirubinemia] who must have a total bilirubin of ≤ 3* ULN) and both AST and ALT < 2.0* ULN
   * For SKd and SMd: Total bilirubin < 2x ULN (except patients with Gilbert's syndrome [hereditary indirect hyperbilirubinemia] who must have a total bilirubin of ≤ 3x ULN) and both AST and ALT < 3.0x ULN
9. Adequate renal function within 28 days prior to C1D1. For Arms 1-11, estimated creatinine clearance (CrCl) calculated using the formula of Cockroft and Gault (1976).

   * ≥ 20 milliliter per minute (mL/min) for SVd, SDd, and SKd arms
   * ≥ 30 mL/min for SNd, SBd, and SMd arms
   * ≥ 45 mL/min for SPd, SPVd, SPEd and SDPd arms
   * > 60 mL/min for SRd arm
10. Adequate hematopoietic function within 28 days prior to C1D1: absolute neutrophil count (ANC) ≥ 1,000/mm^3, hemoglobin (Hb) ≥ 8.0 g/dL, and platelet count ≥ 100,000/mm^3.

    * SPVd (Arm 4) and SKd (Arm 6) only: platelet count ≥150,000.
    * SMd (Arm 12) only: platelet count ≥75,000 for subjects in whom <50% of bone marrow nucleated cells are plasma cells; or platelet count <50,000 for subjects in whom ≥50% of bone marrow nucleated cells are plasma cells.
11. Female patients of childbearing potential must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients must use highly effective methods of contraception throughout the study and for 90 days following the last dose of study treatment. For Arm 12 (SMd), all study subjects must agree and adhere to all testing and contraception requirements as specified in the mezigdomide Global Pregnancy Prevention Plan (PPP)

    SPd (Arm 1) Only.
12. Relapsed or refractory MM with:

    1. Documented evidence of progressive disease (PD) after achieving at least stable disease (SD) for ≥ 1 cycle during a previous MM regimen (i.e., relapsed MM)
    2. ≤ 25 percent (%) response (i.e., patients never achieved ≥ MR) or PD during or within 60 days from the end of the most recent MM regimen (i.e., refractory MM)
    3. Previously undergone ≥ 2 cycles of lenalidomide and a PI (in separate therapeutic regimens [not for maintenance] or in combination)
    4. In the expansion arm at RP2D, patients must not be pomalidomide refractory

    SVd (Arm 2) Only:
13. Relapsed or refractory MM with:

    1. Documented evidence of relapse after ≥ 1 previous line of therapy
    2. Not refractory to bortezomib in their most recent line of therapy

    SRd in RRMM (Arm 3) Only:
14. Patients who received ≥ 1 prior therapeutic regimen (prior lenalidomide is allowed as long as patient's MM was not refractory to prior lenalidomide; patients whose MM was refractory to lenalidomide maintenance regimens will be allowed in this cohort).

    SPVd (Arm 4) Only:
15. Patients who received 1- 3 prior lines of therapy, including ≥ 2 cycles of lenalidomide and have demonstrated disease progression on their last therapy (may include prior bortezomib, as long as the patient's MM was not refractory to bortezomib therapy), but patients must be pomalidomide-naïve in the Dose Expansion at RP2D (Cohort 4.3 ONLY).

    SDd (Arm 5) Only:
16. Patients who received ≥ 3 prior lines of therapy, including a PI and an immunomodulatory agent (IMiD), or patients with MM refractory to both a PI and an IMiD.
17. Patients must not have received prior anti-cluster of differentiation 38 (anti-CD38) monoclonal antibodies (Cohort 5.3 ONLY - Dose Expansion at RP2D).

    SKd (Arm 6) Only:
18. Patients may have received prior PIs; however, their MM must NOT be refractory to carfilzomib.

    SRd in NDMM (Arm 7) Only:
19. Patients must have symptomatic myeloma per IMWG guidelines with either CRAB criteria (calcium elevation, renal failure, anemia, lytic bone lesions) or myeloma-defining events and need systemic therapy. No prior systemic therapy for NDMM is permitted other than pulse dose dexamethasone (maximum dose of 160 mg) or corticosteroid equivalent.

    SNd (Arm 8) Only:
20. Patients must have MM that relapsed after 1 - 3 prior lines of therapy (may not include those with MM refractory to bortezomib or carfilzomib but patients must be ixazomib-naïve).

    SPEd (Arm 9) Only:
21. Patients who received ≥ 2 prior therapies, including lenalidomide and a proteasome inhibitor (in separate or the same regimens), but patients must be pomalidomide-naive and elotuzumab-naive in the Dose Expansion at RP2D (Cohort 9.3 ONLY).

    SBd (Arm 10) Only:
22. Patients who have MM that was refractory to an IMiD, a proteasome inhibitor, and refractory or intolerant (or both) to an anti-CD38 monoclonal antibody. Patients must be belantamab mafodotin-naive in the Dose Expansion cohort at RP2D (Cohort 10.3 ONLY).

    SDPd (Arm 11) Only:
23. Patients who received 1-3 prior therapies, including lenalidomide and a proteasome inhibitor (in separate or the same regimen), but patients must be pomalidomide-naive and daratumumab-naive in the Dose Expansion cohort at RP2D (Cohort 11.3 ONLY).

    SMd (Arm 12) only:
24. Patients with RRMM who have received at least 2 prior lines of therapy, including an IMiD, a PI, and an anti-CD38 monoclonal antibody. Patients must have either failed a T-cell redirecting treatment (eg, CAR-T or bispecific antibody) or otherwise cannot receive such therapy due to either medical or logistic reasons.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not eligible to enroll in this study:

1. Smoldering MM.
2. MM that does not express M-protein or FLC (i.e., non-secretory MM is excluded), and quantitative immunoglobulin levels cannot be used instead.
3. Documented active systemic amyloid light chain amyloidosis.
4. Active plasma cell leukemia.
5. Red Blood Cell (RBC) and platelet transfusions and blood growth factors within 14 days of C1D1 (Arms 1-11 only). Red blood cells and platelet transfusions and blood growth factors within 7 days of C1D1 (Arm 12).
6. Platelet transfusion or G-CSF within 7 days or pegfilgastrim within 14 days prior to the complete blood count (CBC) used to determine eligibility.
7. Radiation, chemotherapy, or immunotherapy or any other tumor-directed therapy ≤ 2 weeks prior to C1D1, and radio-immunotherapy within 6 weeks prior to C1D1. Patients on long-term glucocorticoids during Screening do not require a washout period. Spot radiation is permitted at any time for treatment of fractures or to prevent fractures as well as for pain management.
8. Patients with history of spinal cord compression with residual paraplegia (Dose Escalation Phase only).
9. Treatment with an investigational anti-cancer therapy within 3 weeks prior to C1D1.
10. Prior autologous stem cell transplantation < 1 month, or allogeneic stem cell transplantation < 3 months prior to C1D1.
11. Active graft versus host disease after allogeneic stem cell transplantation.
12. Life expectancy < 3 months.
13. Major surgery within 4 weeks prior to C1D1.
14. Active, unstable cardiovascular function:

    1. Symptomatic ischemia, or
    2. Uncontrolled clinically-significant conduction abnormalities (e.g., patients with ventricular tachycardia on antiarrhythmics are excluded; patients with 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) will not be excluded), or
    3. Congestive heart failure (CHF) of New York Heart Association (NYHA) Class ≥ 3, or
    4. Myocardial infarction (MI) within 3 months prior to C1D1
    5. Ejection fraction (EF) < 50% at Screening (Arms 1-11 only, screening echocardiogram not required for Arm 12, SMd)
15. Uncontrolled active hypertension (Arms 1-11 only).
16. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose.
17. Known active hepatitis A, B or C.
18. Known human immunodeficiency virus (HIV) infection or HIV seropositivity.
19. Any active gastrointestinal dysfunction that prevents the patient from swallowing tablets or interferes with absorption of study treatment.
20. Currently pregnant or breastfeeding.
21. A serious active psychiatric or active medical condition which, in the opinion of the Investigator, could interfere with treatment.
22. Hypersensitivity to any of the treatments for the arm in which the patient is enrolled.
23. SVd Arm (Arm 2), SPVd (Arm 4), and SNd Arm (Arm 8) only: Prior history of neuropathy Grade > 2, or Grade ≥ 2 neuropathy with pain at Screening (within 28 days prior to C1D1).
24. Patients who are eligible for the selinexor PK Run-in only: Treatment with moderate or strong inhibitors/inducers of CYP3A within 7 days prior to Day 1 of the PK Run-in period.
25. Patients who are eligible for the selinexor PK Run-in only: Not able to receive a strong CYP3A4 inhibitor due to concomitant medications.
26. SKd arm only: HBs Ag + plus HBc Ab + even though no active hepatitis B virus (HBV) hepatitis. If HBs Ag - plus HBc Ab +, treating physician needs to contact the medical monitor.
27. Prior exposure to a selective inhibitor of nuclear export (SINE) compound, including selinexor.

    SBd (Arm 10): Only:
28. Current corneal epithelial disease except mild punctate keratopathy.

    SMd (Arm 12 only):
29. History of allogeneic stem cell or solid organ transplant at any time.
30. History of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, pomalidomide (including ≥Grade 3 rash during prior thalidomide, lenalidomide, or pomalidomide therapy), carfilzomib or dexamethasone, any CELMoD agents, or the excipients contained in the formulations, or subject has any contraindications per local prescribing information.
31. Subject is unable or unwilling to agree to refrain from donating blood while on study intervention, during dose interruptions, and for at least 28 days following the last dose of study intervention.
32. Subject is unable or unwilling to undergo protocol required thromboembolism prophylaxis.
33. Use of strong CYP3A4 modulator or proton-pump inhibitors (eg, omeprazole, lansoprazole), within 2 weeks of starting study intervention.
34. Active concomitant malignancies or history of another malignancy within 3 years prior to C1D1 except for adequately treated early-stage basal cell or squamous cell carcinoma of skin, adequately treated carcinoma in situ of breast or cervix, or organ confined prostate cancer.
35. History of chronic hepatitis B with detectable viral load.
36. Subject is unable or unwilling to receive protocol-required dual antiemetic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (Dose-escalation): Maximum Tolerated Dose (MTD) | 12 months
  MTD for once weekly and twice weekly selinexor dose cohorts in the 11 Arms will be evaluated.
Phase 1 (Dose-escalation): Recommended Phase-2 dose (RP2D) | 12 months
  RP2D for each Arm will be determined.
Phase 1 (Dose-escalation): Maximum Plasma Concentration (Cmax) of Selinexor | Pre-dose, 1 hour, 1.5, 2, 3, 4, 5, 6, 8, and 24 hours post-dose on Day 1 (without clarithromycin) and Day 8 (with clarithromycin)
  Cmax of selinexor over a dosing interval when given with and without clarithromycin.
Phase 1 (Dose-escalation): Area Under the Concentration-time Curve From Time Zero to the Last Non-zero Concentration (AUC0-t) of Selinexor | Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 8, and 24 hours post-dose on Day 1 (without clarithromycin) and Day 8 (with clarithromycin)
  Total exposure of selinexor in the blood (AUC0-last) from the time of dosing to the last measurable concentration collected when given with and without clarithromycin.
Phase 1 (Dose-escalation): Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated) (AUC0-inf) | Pre-dose, 1, 1.5, 2, 3, 4, 5, 6, 8, and 24 hours post-dose on Day 1 (without clarithromycin) and Day 8 (with clarithromycin)
Phase 2 (Expansion): Overall response rate (ORR) | 12 months
  ORR for each Arm independently. ORR to include stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR), according to the International Myeloma Working Group (IMWG) criteria.
Phase 2 (Expansion): Duration of response (DOR) | 12 months
  Duration of response for each Arm. DOR is defined as the number of days from the date of the first evidence of objective response until progression.
Phase 2 (Expansion): Clinical Benefit Rate (CBR) | 12 months
  CBR is defined the point estimate of the percentage of patients in that arm who have a response of sCR, CR, VGPR, PR or Minimal response (MR), as assessed by IMWG criteria.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (16):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Jonnsson Comprehensive Cancer Center / University of Los Angeles, Los Angeles, California
  - Sarah Cannon-Colorado Blood Cancer Institute, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - Columbia University, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Wilmot Cancer Center/ University of Rochester, Rochester, New York
  - University of North Carolina - Chapel Hill Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke Institute of Cancer/ Duke University, Durham, North Carolina
  - Sarah Cannon- Tennessee Oncology Nashville, Nashville, Tennessee
  - Fred Hutch Cancer Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- Canada (9):
  - Tom Baker Cancer Center/Alberta Health Services, Calgary, Alberta
  - Cross Cancer Institute / University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Memorial Hospital of Newfoundland, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Royal Victoria Hospital / McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] White D, Schiller GJ, Madan S, Lentzsch S, Chubar E, Lavi N, Van Domelen DR, Bentur OS, Baljevic M. Efficacy and safety of once weekly selinexor 40 mg versus 60 mg with pomalidomide and dexamethasone in relapsed and/or refractory multiple myeloma. Front Oncol. 2024 May 17;14:1352281. doi: 10.3389/fonc.2024.1352281. eCollection 2024. PMID 38826786
- [Derived] Schiller GJ, Lipe BC, Bahlis NJ, Tuchman SA, Bensinger WI, Sutherland HJ, Lentzsch S, Baljevic M, White D, Kotb R, Chen CI, Rossi A, Biran N, LeBlanc R, Grosicki S, Martelli M, Gunsilius E, Spicka I, Stevens DA, Facon T, Mesa MG, Zhang C, Van Domelen DR, Bentur OS, Gasparetto C. Selinexor-Based Triplet Regimens in Patients With Multiple Myeloma Previously Treated With Anti-CD38 Monoclonal Antibodies. Clin Lymphoma Myeloma Leuk. 2023 Sep;23(9):e286-e296.e4. doi: 10.1016/j.clml.2023.06.001. Epub 2023 Jun 5. PMID 37393120
- [Derived] Bahlis NJ, Sutherland H, White D, Sebag M, Lentzsch S, Kotb R, Venner CP, Gasparetto C, Del Col A, Neri P, Reece D, Kauffman M, Shacham S, Unger TJ, Jeha J, Saint-Martin JR, Shah J, Chen C. Selinexor plus low-dose bortezomib and dexamethasone for patients with relapsed or refractory multiple myeloma. Blood. 2018 Dec 13;132(24):2546-2554. doi: 10.1182/blood-2018-06-858852. Epub 2018 Oct 23. PMID 30352784